CLINICAL TRIAL: NCT06421155
Title: A Pilot Study of Brain Magnetic Resonance Fingerprinting in Children, Adolescents and Young Adults With Acute Leukemia
Brief Title: Brain MRF in Children, Adolescents and Young Adults With Acute Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE3923
Record Dates: First submitted 2024-04-30; First posted 2024-05-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Leukemia; Acute Lymphoblastic Leukemia, Pediatric; Acute Myeloid Leukemia in Children; Myeloproliferative Neoplasm
Keywords: Acute Leukemia Children; Acute Leukemia Adolescents; Acute Leukemia Young Adults
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRF +/-Neurocognitive Testing (Other): Once the participants meeting the inclusion criteria are identified and formally consent to participate in the study, each participant will undergo a baseline MRF imaging exam along with the neurocognative testing, preferably prior to starting induction chemotherapy. The total treatment duration for an individual participant can vary anywhere between 6 months - 3 years depending on the type of acute leukemia, so investigator plans to obtain MRF scans every 6 months during the therapy as well as during the first year of the off -therapy period
  Interventions: Other: MRF with neurocognative studies

INTERVENTIONS:
Other: MRF with neurocognative studies — Magnetic Resonance Imaging is used to assess the risk of neurocognitive side effects in pediatric and AYA patients with acute leukemia receiving chemotherapy and participants will also be asked to complete a neurocognitive battery designed by Cogstate and administered on iPad in a simple gaming format

SUMMARY:
The survival of children, adolescents and young adults (AYA) with acute leukemia has improved dramatically over the last two decades. This success is a result of using multiple chemotherapy drugs in combination, with the inclusion of drugs that enter the brain and prevent leukemia cells from growing there. Studies in these cancer survivors have shown that the exposure to these chemotherapy drugs can lead to risks for impaired brain function, also referred to as neurocognitive side effects of chemotherapy. There is an opportunity to identify participants at risk for these side effects and to prevent their development. The purpose of this study is to incorporate a brain imaging tool known as Magnetic Resonance Fingerprinting (MRF) to look for brain matter changes in acute leukemia participants receiving chemotherapy. The MRF scan will be performed at diagnosis and repeated at multiple times during the entire therapy duration as well as at defined intervals after therapy is complete. Investigators would also do an electronic test of memory and brain function (cognitive function), which would be administered in a gaming format on iPads or a similar device. The goal will be to correlate results of MRF imaging with the tests of cognitive function. The benefits of this imaging technique include that it can be done quickly (in minutes), it is non-invasive, it is resistant to motion-artifacts and it can be easily repeated for comparison purposes. The advantages of the cognitive test include its short duration of 20 minutes and its gaming format making it friendly for children to use.

DETAILED DESCRIPTION:
Acute leukemia (AL), including Acute Lymphoblastic Leukemia (ALL), Acute Myeloid Leukemia (AML) and myeloproliferative neoplasms (MPN) are among the most common childhood cancers, the 5-year overall survival of children with leukemia has significantly improved with the current treatment methods, and is now ~90 % for ALL participants and ~70 % for AML participants. There has been a remarkable shift in the treatment strategy for childhood acute leukemia to reduce the burden of therapy related complications. Most notably, the addition of central nervous system (CNS)-directed, intensified intravenous and intrathecal chemotherapy regimens for most standard risk participants has obviated the need for craniospinal radiation therapy (CRT), thus reserving CRT for high-risk participants. With the improved overall survival rates, there is an increasing focus on characterizing and mitigating the long-term effects of the disease and therapy that may affect the quality of life of these participants. The results of multiple studies have indicated that the long-term survivors of ALL and AML experience varying degrees of neurocognitive deficits including memory loss, poor concentration, deficits in executive functioning and personality changes5-9. Methotrexate which is an important chemotherapeutic agent in the treatment of acute leukemia is known to cause chemotherapy induced cognitive impairment (CICI), by causing complex glial dysfunction leading to disruption of activity-dependent myelination in the CNS.

Studies designed to characterize normal brain development in early childhood have not only contributed significantly to our understanding of healthy neurodevelopment, but have also helped to identify neurodevelopmental problems at an early stage, enabling the application of treatment interventions in a timely fashion. Although magnetic resonance imaging (MRI) has been used for this purpose, its application has been hampered by several limitations including the sensitivity to motion artifact, the length of time required to perform a scan, and the requirement for sedation for younger participants. These limitations can be overcome using a new technology known as magnetic resonance fingerprinting (MRF), which allows for rapid, efficient and simultaneous quantification of multiple tissue properties, and quantifies T1, T2 and Myelin Water Fraction (MWF) simultaneously. Sedation is not necessary since whole brain MRF imaging takes approximately 5 minutes to complete and is resistant to motion artifacts.

These properties position MRF for use to assess multiple tissue properties in both pediatric and AYA participants diagnosed with acute leukemia, before, during and after exposure to CNS directed chemotherapy. The investigator proposes to use MRF to monitor demyelination, which has been documented as an underlying mechanism contributing to the long-term neurocognitive deficits seen in participantsundergoing chemotherapy. The goal of using MRF in this context is that it might ultimately serve as a valuable imaging biomarker that would enable early detection of the participants that are at an increased risk of developing neurocognitive deficits due to exposure to anti-neoplastic chemotherapy, by detecting the myelin changes as defined by MRF quantification of myelin water fraction. The capacity for detection would facilitate development of early interventions for these high-risk participants, so that their quality of life can be preserved as much as possible.

The study will evaluate the feasibility of obtaining MRF imaging data along with assessments of neurocognitive function. Chanages/decline in neurocognitive function in pediatric participants undergoing treatment for acute leukemia have been tested, validated and reported by the Children's Oncology Group using a battery of assessment developed by Cogstate®. The computerized cognitive tests are rapid, reliable, and have demonstrated sensitivity to drug related changes in cognition. The tests have been designed and validated to withstand operational challenges during the conduction of clinical trials. The data system is HIPAA compliant U.S. FDA Class II Exempt Digital Medical Device.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 0 - 30 years
* Participants from University Hospitals Rainbow Babies & Children's Hospital, UH Seidman Cancer Center, and participants referred from outside facilities diagnosed with acute leukemia.
* Meets diagnostic criteria for acute leukemia including acute lymphocytic leukemia (ALL), acute myeloid leukemia (AML) and myeloproliferative neoplasm/leukemia.
* Participants must have the ability to understand and the willingness to sign a written informed consent document. Participants who are 14 years and older must have the ability to understand and the willingness to sign a written informed consent document. Participants who are between the ages of 7 to 13 will be given an information sheet that explains the study to them. The information sheet may be used for study participants between the ages of 14-17 if it would better inform the child about the nature and procedures that will undergo as a participant in the study.

Exclusion Criteria:

* Individuals that are >2 weeks into the induction chemotherapy for acute leukemia.
* Individuals with either a heart pacemaker, heart defibrillator, metal in the eye, some types of metal elsewhere within the body such as certain surgical clips for aneurysms in the head, heart valve prostheses, electrodes, some other implanted devices, or any other MRI contraindication

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2028-06-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of alterations in brain structure as measured by mean myelin water fraction | Baseline and during chemotherapy(up to 3.5 years)
  Mean myelin water fraction is measured by Student's T-test. The two-tailed means comparison will be considered statistically significant if a p-value of less than 0.5 is observed.

SECONDARY OUTCOMES:
Incidence of change in tissue evaluation using brain property mapping | Baseline, every 6 months during the duration of therapy(up to 3.5 years), and every 6 months during the first year of the off-therapy period.
  Brain tissue property maps assessed using MRF scans

OTHER OUTCOMES:
Incidence of brain tissue changes using neurocognitive testing | Baseline, every 6 months during the duration of therapy(up to 3.5 years), and every 6 months during the first year of the off-therapy period.
  Cognitive assessment using Cogstate software

CONTACTS AND LOCATIONS:
Overall Officials: Mari Dallas, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Rainbow Babies & Children's Hospital, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Rainbow Babies & Children's Hospital, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical diagnosis, treatment, MRI/MRF and neurocognitive testing
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be provided within 12 months from study completion and for at least 6 years after study closure.
Access Criteria: Study team will only have access to submit data